CLINICAL TRIAL: NCT03756259
Title: Understanding the Reasons for Delay in Seeking Care for Pneumonia and Recurrent Wheeze Among Caregivers of Children Under Five in Pakistan
Brief Title: Pneumonia Perception Project-Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AC 18109
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2019-05

CONDITIONS: Pneumonia; Perception, Self
MeSH Terms: conditions — Pneumonia | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pneumonia perception arm (Other): Caregivers of children under five will be interviewed qualitatively to understand in depth on perception of pneumonia. These will be mothers, fathers and grandmothers of these children. Once the formative research is done, it will inform design of an intervention whereby the caregivers will be recruited to be counselled by Lady health workers on pneumonia and its prevention via an audiovisual user friendly android based mobile application. Additionally, one text and one voice message will also be sent to the caregivers cell phones on the same subject. The LHWs will also be trained on pneumonia case finding which they will manage at their end and refer if required while doing daily field visits.
  Interventions: Behavioral: Mobile Health (mHealth) for Pneumonia

INTERVENTIONS:
Behavioral: Mobile Health (mHealth) for Pneumonia — Audiovisual mobile based application will be used to counsel caregivers of children under five on pneumonia and its prevention. This will be coupled with text and voice message dissemination to the cell phones of caregivers and active pneumonia case finding by the LHWs which will be managed according to severity.

SUMMARY:
Pneumonia and recurrent wheeze contribute extensively to under five childhood morbidity and mortality in Pakistan. Among the avoidable causes of death due to these diseases, delayed care seeking is a major one whereby around 38% of deaths due to acute respiratory illnesses occur in households. Of these cases which die due to delayed care seeking, majority are taken for healthcare after 2 days of initiation of symptoms with around 30% been given antibiotics at home before seeking healthcare. Around 32% of these cases die at home, 48% in hospitals, 9% en route, and the 11% in clinics or health centres.This could be due to lack of time, lack of funds for healthcare, lack of decision making on the part of the mother or improper carer perception of the seriousness of the condition. Thus there are various cultural, social, personal and religious factors which affect the care seeking behaviors of caregivers for these illnesses. Understanding these aspects of delayed care seeking is critical to develop effective intervention strategies to reduce disease related mortality. We, therefore, aim to establish an understanding of perception of under-five pneumonia and recurrent wheeze among caregivers of children under five along with associated factors of delayed care seeking in selected communities in Pakistan. The results of this study will permit us to design an effectiveness study which can be used by program managers and policy makers to develop program strategies to reduce childhood deaths due to delayed care seeking for these diseases.

DETAILED DESCRIPTION:
Background: In Pakistan, pneumonia and recurrent wheeze in children under five pose significant threats to children's health. Despite being preventable, more than 90,000 children die each year due to pneumonia in Pakistan, making it one of the top five countries in the world, with the highest pneumonia related childhood mortality. Similarly, children account for 20%-30% of the 2 million Pakistani asthma patients. The predisposing factors which lead to these illnesses include lack of hygiene, lack of immunization, overcrowding, household air pollution, smoking and poverty. Prompt recognition and timely initiation of treatment is imperative in children under five with pneumonia and recurrent wheeze and failure to do so can lead to complications and death.

In children under five, among the causes of death due to these diseases, one is delayed care seeking. It has been identified that around 38% of deaths due to respiratory illnesses occur in households due to this delayed care seeking which is defined as delay in care sought for an illness outside home. This delay is referred to as the time taken by the caregiver to seek healthcare later than what would have been optimal.

In most of the Low middle income countries (LMICs), carer gender plays an important role in decisions to seek care. Although in majority of households, the primary caregivers of children under five are the mothers of those children, decisions with respect to care are often made by fathers or mothers in law which is a problem as they do not cater to the child in a timely manner either by not being there or being ignorant of basic management of the illness. Another contributing factor could be lack of time to take the child for healthcare as the mothers are usually occupied in their household chores and the fathers are busy working. And in rare cases where either the mother of a child dies at childbirth (500 per 100,000 live births) and when fathers are working away from home, it is the secondary caregiver who is responsible for care-seeking of that child. He/she could be an aunt/uncle or neighbour. But in such cases often the child is neglected due to other priorities of the secondary caregivers.

Although well-proven life-saving tools are available to stop mortality due to preventable illnesses like pneumonia and recurrent wheeze, the existing health systems in Pakistan are passive. Here, healthcare providers tend to wait for patients to come to them but the later the patients with acute respiratory illness come, the more likely they are to die. World Health Organization (WHO) and United Nations International Children's Emergency Fund (UNICEF) have, therefore, emphasized the development of innovative, sustainable and cost-effective strategies/interventions to improve child health. It is important to devise a strategy whereby patient's symptoms are identified timely and immediate care given at their doorstep. Experimental studies provide the strongest evidence that illness perceptions can modify behaviours and care-seeking, and several studies have shown that interventions designed to change illness perceptions can improve health outcomes. Locally adapted behaviour change communication may reduce the incidence of severe pneumonia and could be a key component in national child-health strategies.

One of the most impactful strategies can be timely healthcare seeking through community health workers who have been a powerful force to promote healthy behaviours and extend the reach to the health system by acting as a bridge between the community and the system. Community-based packaged interventions delivered through CHWs have been shown to improve care seeking for childhood illnesses. In Pakistan, these CHWs are referred to as Lady Health Workers (LHWs) enrolled under the National Program for Family Planning and Primary Healthcare. On average each LHW covers 100-150 households by making monthly visits and providing basic health services and education on health and wellbeing. These LHWs could, therefore, be a useful mode of active pneumonia and recurrent wheeze case finding and information sharing to counsel against development of acute respiratory infections as evidence has shown that health interventions integrating Community Health Workers (CHWs) can lead to positive behaviour changes and lower morbidity and mortality rates, while moving services and information closer to the communities where they are actually needed.

Objective: Our study will explore healthcare care-seeking for childhood pneumonia and recurrent wheeze among caregivers of children under five through a qualitative approach. Further, we aim to devise a Care Model to actively find cases through LHWs and promote appropriate care seeking behaviour among the caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children under five
* Those consenting to participate

Exclusion Criteria:

* Children with any long standing chronic illness

Ages: 1 Minute to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of perception of caregivers of children under five on pneumonia and recurrent wheeze | 6 months
  The qualitative approach will provide a detailed understanding of perception of pneumonia and recurrent wheeze among caregivers of children under five
Improvement in perception of pneumonia and recurrent wheeze among caregivers of children under five | 6 months
  Through the mobile based intervention we plan to improve caregiver perception on pneumonia and recurrent wheeze
Active case finding of pneumonia by lady health workers | 6 months
  LHWs will identify pneumonia cases and manage or refer them as the case may be

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- MNCHRN, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No